CLINICAL TRIAL: NCT05877365
Title: Effects of Standard Process's 21-day Guided Purification Program on Metabolic Health in College Setting
Brief Title: Effects of 21-day Purification Program on Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Standard Process Inc. (Industry)
Collaborators: Keiser University College of Chiropractic Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: SP-019-2
Record Dates: First submitted 2023-03-10; First posted 2023-05-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy
Keywords: Purification; Whole Food Vitamins; Detoxification

STUDY DESIGN:
Intervention Model Description: diet only vs whole food supplement based intervention
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Only (No Intervention): Following the same diet as the Purification group
- Purification (Experimental): Following a diet along with whole food based supplementation
  Interventions: Dietary Supplement: Standard Process 21-Day Purification Program

INTERVENTIONS:
Dietary Supplement: Standard Process 21-Day Purification Program — Purification, also known as detoxification, may help remove natural toxins from the body, while maintaining a healthy weight. The toxin load humans are exposed to daily may take a toll on physical and emotional well-being. Internally, human bodies produce waste byproducts because of normal metabolic function. Although the body is designed to rid itself of these toxins naturally, it can become overburdened. Purification may offer the body additional support to expel these toxins and manage weight, which is important to maintaining health and vitality.
  Arms: Purification

SUMMARY:
This is a study to assess the impact of Standard Process's 21-Day Purification Program on metabolic health. Participants will be given the opportunity to consume the complex combination of vitamins, minerals, and antioxidants that comprise the 21-Day Guided Purification Program by Standard Process.

DETAILED DESCRIPTION:
Purification, also known as detoxification, may help remove natural toxins from the body, while maintaining a healthy weight. The toxin load we are exposed to daily may take a toll on our physical and emotional well-being. Internally, human bodies produce waste byproducts because of normal metabolic function. Although the human body is designed to rid itself of these toxins naturally, it can become overburdened. Purification may offer the body additional support to expel these toxins and manage weight, which is important to maintaining health and vitality.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee.
* Willingness to comply with study protocol for 58 days
* Willingness to come and provide samples on all 4 study visits
* No allergy to any study products (a complete list of what supplements will assist is provided below))
* Subject is >18 years of age
* Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit, and is not actively planning a pregnancy
* If on a chronic medication (that does not result in exclusion), subject has been on stable dose for at least two months prior to screening visit
* Subject has at least two weeks wash out period between completion of a previous research study that required ingestion of any study food or drug and their start in the current study
* Willingness to stay compliant for 22 days and not participate in another research study

Exclusion Criteria:

* Prohibited Medications, Supplements or Herbal Products

  * Subjects who are experiencing any adverse events due to any nutraceutical, OTC, or pharmaceutical or investigational products
  * Celiac and other gastrointestinal health concerns
  * Subjects may not receive any other investigational products not part of normal clinical care
  * Lipid lowering drugs in the preceding 4 weeks and for duration of study [examples- statins, cholesterol absorption inhibitors like Ezetimibe (Zetia), PCSK9 inhibitors like Alirocumab (Praluent), Evolocumab (Repatha) etc.]
  * The use of anticoagulant medications in the preceding 4 weeks and for duration of study [Examples: apixaban (Eliquis), betrixaban (Bevyxxa), edoxaban (Savaysa), and rivaroxaban (Xarelto) etc.]
* Pregnant and nursing women are excluded from participation and women of childbearing age expecting to be pregnant soon will be excluded from the study
* Subjects with untreated endocrine, neurological, or infectious disease
* Subjects with the diagnosis of HIV disease or AIDS
* Significant liver or kidney disease (recent or ongoing hepatitis, cirrhosis, glomerulonephritis, dialysis treatment)
* Rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematosus, polymyositis, scleroderma, polymyalgia rheumatic, temporal arteritis or Reiter's Syndrome
* Psoriasis, Deep vein thrombosis or pulmonary embolus (blood clot to lungs)
* History of cancer
* Serious medical illness like high TG levels >150 mg/DL for example
* Substance Use - Use of ethanol within 24 hours of the evaluation visits (all 4 visits)
* Any other sound medical, psychiatric and/or social reason as determined by the PI
* Co-enrollment in other studies is restricted. Study staff should be notified of co-enrollment as it may require the approval of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Porphyrins in Urine | 58 days
  Using a kit, urinary porphyrins will be measured.

SECONDARY OUTCOMES:
Changes in GGT | 58 days
  A blood draw will be performed to evaluate gamma-glutamyl transferase (GGT) levels
Changes in GST | 58 days
  A blood draw will be performed to evaluate Glutathione S-Transferase (GST) levels
Questionnaire | 58 days
  PROMIS Global 10 Health Questionnaire will be used for the participant to evaluate their own health on a scale from 1-5.
Changes in Weight | 58 days
  Participants will be weighed at each visit to help evaluate health

CONTACTS AND LOCATIONS:
Overall Officials: Chinmayee Panda, PhD, Principal Investigator — Standard Process Inc.
Locations (1):
- Keiser University Spine Care Clinic, West Palm Beach, Florida, United States

REFERENCES:
- [Background] Sears ME, Genuis SJ. Environmental determinants of chronic disease and medical approaches: recognition, avoidance, supportive therapy, and detoxification. J Environ Public Health. 2012;2012:356798. doi: 10.1155/2012/356798. Epub 2012 Jan 19. PMID 22315626
- [Background] Liska DJ. The detoxification enzyme systems. Altern Med Rev. 1998 Jun;3(3):187-98. PMID 9630736
- [Background] Liska D, Lyon M, Jones DS. Detoxification and biotransformational imbalances. Explore (NY). 2006 Mar;2(2):122-40. doi: 10.1016/j.explore.2005.12.009. No abstract available. PMID 16781626
- [Background] Hodges RE, Minich DM. Modulation of Metabolic Detoxification Pathways Using Foods and Food-Derived Components: A Scientific Review with Clinical Application. J Nutr Metab. 2015;2015:760689. doi: 10.1155/2015/760689. Epub 2015 Jun 16. PMID 26167297
- [Background] Griendling KK, Touyz RM, Zweier JL, Dikalov S, Chilian W, Chen YR, Harrison DG, Bhatnagar A; American Heart Association Council on Basic Cardiovascular Sciences. Measurement of Reactive Oxygen Species, Reactive Nitrogen Species, and Redox-Dependent Signaling in the Cardiovascular System: A Scientific Statement From the American Heart Association. Circ Res. 2016 Aug 19;119(5):e39-75. doi: 10.1161/RES.0000000000000110. Epub 2016 Jul 14. PMID 27418630
- [Background] Zweier JL, Duke SS, Kuppusamy P, Sylvester JT, Gabrielson EW. Electron paramagnetic resonance evidence that cellular oxygen toxicity is caused by the generation of superoxide and hydroxyl free radicals. FEBS Lett. 1989 Jul 31;252(1-2):12-6. doi: 10.1016/0014-5793(89)80881-6. PMID 2547649
- [Background] Pastore A, Federici G, Bertini E, Piemonte F. Analysis of glutathione: implication in redox and detoxification. Clin Chim Acta. 2003 Jul 1;333(1):19-39. doi: 10.1016/s0009-8981(03)00200-6. PMID 12809732
- [Background] Lee DH, Blomhoff R, Jacobs DR Jr. Is serum gamma glutamyltransferase a marker of oxidative stress? Free Radic Res. 2004 Jun;38(6):535-9. doi: 10.1080/10715760410001694026. PMID 15346644
- [Background] Chen CA, Wang TY, Varadharaj S, Reyes LA, Hemann C, Talukder MA, Chen YR, Druhan LJ, Zweier JL. S-glutathionylation uncouples eNOS and regulates its cellular and vascular function. Nature. 2010 Dec 23;468(7327):1115-8. doi: 10.1038/nature09599. PMID 21179168
- [Background] Varadharaj S, Kelly OJ, Khayat RN, Kumar PS, Ahmed N, Zweier JL. Role of Dietary Antioxidants in the Preservation of Vascular Function and the Modulation of Health and Disease. Front Cardiovasc Med. 2017 Nov 1;4:64. doi: 10.3389/fcvm.2017.00064. eCollection 2017. PMID 29164133
- [Background] Kim JA, Kim JY, Kang SW. Effects of the Dietary Detoxification Program on Serum gamma-glutamyltransferase, Anthropometric Data and Metabolic Biomarkers in Adults. J Lifestyle Med. 2016 Sep;6(2):49-57. doi: 10.15280/jlm.2016.6.2.49. Epub 2016 Sep 30. PMID 27924283
- [Background] Brewster MA. Biomarkers of xenobiotic exposures. Ann Clin Lab Sci. 1988 Jul-Aug;18(4):306-17. PMID 3044268
- [Background] Bonakdar RA, Sweeney M, Dalhoumi S, Adair V, Garvey C, Hodge T, Herrala L, Barbee A, Case C, Kearney J, Smith K, Hwang J. Detoxification Enhanced Lifestyle Intervention Targeting Endotoxemia (DELITE) in the Setting of Obesity and Pain: Results of a Pilot Group Intervention. Integr Med (Encinitas). 2020 Oct;19(5):16-28. PMID 33488302
- [Derived] Panda C, Kruse R, Williams K, Nance B, Gudavalli M, Pourafshar S, Metzger B, Komarnytsky S. Metabolic reset purification program improves antioxidant balance and gut microbiome in individuals transitioning to a healthier diet. Front Nutr. 2025 Aug 11;12:1621709. doi: 10.3389/fnut.2025.1621709. eCollection 2025. PMID 40860479